CLINICAL TRIAL: NCT05246345
Title: Venetoclax Resistance Landscape in Chronic Lymphocytic Leukemia
Acronym: RAVEN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 GUIEZE; 2021-A00362-39 (Other: 2021-A00362-39)
Record Dates: First submitted 2021-10-13; First posted 2022-02-18 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-06

CONDITIONS: Chronic Lymphocytic Leukemia; CLL; Progressive Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Relapsed Chronic Lymphocytic Leukemia
Keywords: Venetoclax; Venetoclax resistance; Resistance mechanism
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax: Cohort of refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax

SUMMARY:
The purpose of this study is to collect medical informations and samples from refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax treatment, in order to evaluate the frequency of resistance mechanisms.

DETAILED DESCRIPTION:
The purpose of this study is to collect medical informations and samples (blood, bone marrow and/or lymph node) from refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax treatment, in order to evaluate the frequency of resistance mechanisms (BCL2 mutations, over-expression of other members of the BCL2 protein family and energy metabolism changes).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old;
* chronic lymphocytic leukemia diagnosis according to iwCLL criteria;
* refractory and/or relapsed disease during or after venetoclax treatment;
* tumor samples available.
* Relapse might be progressive chronic lymphocytic leukemia or transformation into Richter syndrome.
* Patients must be able to express their opposition to be enrolled in this study, if need be.
* Patients must be affiliated at the French Social Security system

Exclusion Criteria:

Patients of their legal guardians refusing to participate

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lymphocytic leukemia diagnosis according to iwCLL criteria and who are refractory and/or relapsed disease during or after venetoclax treatment; tumor samples available.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Frequency measurement of BCL2 gene mutations | immediately after the chronic lymphocytic leukemia progression
  Frequency measurement of BCL2 gene mutations in a cohort of refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax therapy

SECONDARY OUTCOMES:
Frequency measurement of 1q amplification | immediately after the chronic lymphocytic leukemia progression
  Frequency measurement of 1q amplification in a cohort of refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax therapy
Differential expression of candidate transcripts and proteins | immediately after the chronic lymphocytic leukemia progression
  Differential expression of candidate transcripts and proteins (BCL2 protein family, AMP signaling pathway, energy metabolism) in a cohort of refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax therapy
Correlation of resistance mechanisms with clinical staging | immediately after the chronic lymphocytic leukemia progression
  Correlation of resistance mechanisms (BCL2 mutation and 1q amplification) with clinical staging, in a cohort of refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax therapy
Correlation of resistance mechanisms with genomic chronic lymphocytic leukemia features | immediately after the chronic lymphocytic leukemia progression
  Correlation of resistance mechanisms (BCL2 mutation and 1q amplification) with genomic chronic lymphocytic leukemia features, in a cohort of refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax therapy
Progression Free Survival according to resistance mechanisms | immediately after the chronic lymphocytic leukemia progression
  Progression Free Survival according to resistance mechanisms (BCL2 mutation and 1q amplification), in a cohort of refractory and/or relapsed chronic lymphocytic leukemia during or after venetoclax therapy

CONTACTS AND LOCATIONS:
Overall Officials: Romain GUIEZE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (14):
- France (14):
  - CHU d'Amiens, Amiens
  - CHU de Besançon, Besançon
  - Hopital AVICENNE, Bobigny
  - CHU clermont-ferrand, Clermont-Ferrand
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Centre LEON BERARD, Lyon
  - CHU de Montpellier, Montpellier
  - CHU Nancy, Nancy
  - Hopital Pitié Salpetrière, Paris
  - Hopital Haut LEVEQUE, Pessac
  - CHU de Reims, Reims
  - IUCT Oncopole, Toulouse